CLINICAL TRIAL: NCT06092151
Title: A Feasibility Study to Determine Whether a Randomised Controlled Trial of Silver Diamine Fluoride Compared to Usual Care for the Management of Caries in Children's Primary Teeth is Feasible in UK Primary Dental Care
Brief Title: SDF for the Management of Dental Caries in Children in Primary Dental Care: Protocol for a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH21666
Record Dates: First submitted 2023-06-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Intervention Model Description: feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Diamine Fluoride (Experimental): SDF treatment for caries in the primary teeth of children included
  Interventions: Device: Silver diamine fluoride
- Usual Care (Active Comparator): Usual care determined by child's dentist for caries in their primary teeth
  Interventions: Procedure: Usual dental care

INTERVENTIONS:
Device: Silver diamine fluoride — silver diamine fluoride - maximum 1 drop to be applied per visit (manufacturer advises this would treat up to 5 teeth)
  Arms: Silver Diamine Fluoride
Procedure: Usual dental care — Usual restorative or preventative care determined by the child's dentist - for examples fillings or crowns
  Arms: Usual Care

SUMMARY:
Dental caries remains a significant health problem in England, effecting 11% of 3-year-olds and 23% of 5-year- olds. Children with dental caries suffer pain, infection and poor oral health-related quality of life. There are different approaches for the management of childhood dental caries but it remains the most common reason for a hospital admission in the UK for children aged 5-9 years, costing the NHS £50 million in 2015-2016. While current approaches have been extensively investigated, their ability to: 1) control pain and infection; 2) prevent hospital admissions, and 3) be implemented within the current NHS contractual arrangements, remains unsatisfactory. Silver diamine fluoride (SDF) is an alternative and non-invasive approach that is applied topically (simple to manage for children) and has proven efficacy in arresting caries progression in primary teeth, principally from studies conducted outside Europe. Its use in primary dental care practice in the UK is limited despite acknowledged need.

However, the clinical and cost effectiveness of SDF has not been compared to usual care in the UK, so it is unknown which treatment is more effective. Before a pragmatic randomised controlled trial (RCT) can be conducted into the clinical and cost effectiveness of SDF compared to usual care, there are several uncertainties related to recruitment, retention and fidelity that require investigation in a feasibility study.

Research Question Is a randomised controlled trial (RCT) to compare the effectiveness of silver diamine fluoride (SDF) to usual care for the treatment of caries in children's primary teeth feasible in UK primary dental care? Aim The overall aim is to establish whether conducting a RCT to compare SDF to usual care for the treatment of caries in children's primary teeth is feasible.

Methods This mixed-method study is a feasibility study with an embedded process evaluation, to compare SDF with usual treatment in primary dental care in the UK. It will be individually randomised, with at least eight dentists, each in a different dental practice and a sample size of 80 participants. There will be ten participants per dentist and equal arm allocation. Follow-up will be for one year. The study will inform whether an RCT is feasible by resolving several key uncertainties. Acceptability and implementation of SDF and the research processes will be explored. Patient and Public Involvement and Engagement (PPIE) representatives will be involved throughout, further informing design including recruitment/retention strategies, participant documentation, analysis, engagement and dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-6 years
* Cavitated dentinal caries in any primary tooth
* No carious involvement of the tooth pulp
* No dental infection secondary to a non-vital tooth
* Parent/carer able to complete consent forms (with the support of an interpreter if necessary)

Exclusion Criteria:

* Allergy to any treatment component
* Caries effecting the pulp
* Infection secondary to a non-vital tooth
* Conditions requiring special considerations for the child's dental management where randomisation would not be appropriate for example a medical history including cardiac defects, oncology, hereditary bleeding, or being immunocompromised.
* Dental anomalies effecting the carious teeth involved: amelogenesis imperfecta, dentinogenesis imperfecta, molar incisor hypomineralisation, abnormal morphology such as double teeth.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Data quality of candidate primary outcome measures - ICDAS | 18 months
  • International Caries Detection and Assessment System (ICDAS) - by measuring percentage of completion and data quality
Data quality of candidate primary outcome measure - pain and infection including PUFA | 18 months
  Occurrence or report of pain or infection and Pulpal involvement, Ulceration, Fistula, Abscess (PUFA) index by measuring percentage of completion and data quality
Data quality of candidate secondary outcome measure; referral to secondary care | 18 months
  Referral to secondary care; measuring percentage of completion and data quality
Data quality of candidate secondary outcome measure; Completion course of treatment | 18 months
  Completion course of treatment; measuring percentage of completion and data
Data quality of candidate secondary outcome measure; number of appointments taken for completion of a course of treatment | 18 months
  The number of appointments taken for completion of a course of treatment; measuring percentage of completion and data quality
Data quality of secondary outcome measure; Adherence to intervention protocol or usual care guidelines. | 18 months
  Adherence to intervention protocol or usual care guidelines. ; measuring percentage of completion and data quality
Data quality of candidate secondary outcome measure; Adverse effect(s). | 18 months
  Adverse effect(s). ; measuring percentage of completion and data quality
Data quality of candidate secondary outcome measure; Appointment length | 18 months
  Appointment length; measuring percentage of completion and data quality
Data quality of candidate secondary outcome measure; • number of units of dental activity claimed | 18 months
  Number of units of dental activity claimed; measuring percentage of completion and data quality
Data quality of candidate secondary outcome measure; child and parental/carer reported experience of treatment | 18 months
  Child and parental/carer reported experience of treatment. measuring percentage of completion and data quality
Data quality of candidate secondary outcome measure; Parental/carer reported oral health-related quality of life; P-CPQ16 | 18 months
  Parental/carer reported oral health-related quality of life; measuring percentage of completion and data quality
Variability of primary outcome measure; ICDAS or pain and infection | 18 months
  This will be calculated once the specific measure has been chosen based on completion rates and data quality, and discussion with the study panel.
  Calculation of the variability of the primary outcome measure that is ultimately chosen for a trial should it be deemed feasible.
recruitment, randomisation and retention rates of child participants | 18 months
  Percentage rates of recruitment, randomisation and retention of child participants
recruitment and retention rates of dental professionals | 18 months
  Percentage rates of recruitment and retention of dental professionals
rate of dentists' adherence to the study protocol (treatment allocation) | 18 months
  Percentage of dentists which adhered to the randomisation determined treatment choice for the child
Data quality and percentage completion rates of cost effectiveness data; cost data completed in case report forms by dental professional | 18 months
  Data quality and percentage completion rates of cost effectiveness data; cost data completed in case report forms (time of appointments, treatment carried out, number of UDAs claimed) by dental professional
Data quality of cost effectiveness data; parental questionnaires | 18 months
  Data quality and percentage completion rates of cost effectiveness data; cost questionnaires completed by parents

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Timms L, Rodd H, Deery C, Brocklehurst P, Marshman Z. Silver diamine fluoride for the management of dental caries in children in primary dental care: protocol for a feasibility study. Pilot Feasibility Stud. 2024 Jun 24;10(1):95. doi: 10.1186/s40814-024-01519-y. PMID 38915111